CLINICAL TRIAL: NCT01621906
Title: Pilot Study of 18F-FLT-PET Imaging of the Brain in Patients With Metastatic Breast Cancer to the Brain Treated With Whole Brain Radiation Therapy With or Without Sorafenib: Comparison With MR Imaging of the Brain
Brief Title: 18F-FLT-PET Imaging of the Brain in Patients With Metastatic Breast Cancer to the Brain Treated With Whole Brain Radiation Therapy With or Without Sorafenib: Comparison With MR Imaging of the Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-039
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Results first posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2021-06

CONDITIONS: Metastatic Breast Cancer to the Brain
Keywords: Breast; brain metastases; 18F-FLT-PET Imaging; FLT(3'DEOXY-3'FLUOROTHYMIDINE); MR Imaging; 12-039
MeSH Terms: conditions — Brain Neoplasms

ARMS (2):
- Cohort 1 (Experimental): Cohort 1 will include the first ten patients treated with WBRT concomitantly with sorafenib (on a separate phase I trial). We will perform a pilot study of serial FLT-PET imaging of the brain at baseline (< 4 weeks prior to initiation of WBRT), up to 7-10 days post-WBRT and 10-12 weeks after WBRT in patients with metastatic breast cancer to the brain (N=20) treated with WBRT with or without sorafenib.
  Interventions: Device: 18F-FLT-PET Imaging
- Cohort 2 (Experimental): Cohort 2 will include patients treated with standard WBRT alone. Patients in both these cohorts will also be assessed with standard non-invasive MRI in addition to [18F] FLT PET at baseline (< 4 weeks of WBRT) and 10-12 weeks after completion of WBRT.
  Interventions: Device: 18F-FLT-PET Imaging

INTERVENTIONS:
Device: 18F-FLT-PET Imaging — All patients will be imaged using FLT-PET scans at baseline (within 4 weeks of initiation of WBRT), 7-10 days after completion of WBRT and then 10-12 weeks after WBRT.
  Patients will also be evaluated with MRI imaging at baseline and then 10-12 weeks after WBRT.
  Patients will be followed with MRI every 3 months (+/- 7 days) for the first year and then every 6 months (+/- 7 days) thereafter which is the standard of care.
  Arms: Cohort 1
Device: 18F-FLT-PET Imaging — All patients will be imaged using FLT-PET scans at baseline (within 4 weeks of initiation of WBRT), 7-10 days after completion of WBRT and then 10-12 weeks after WBRT.
  Patients will also be evaluated with MRI imaging at baseline and then 10-12 weeks after WBRT.
  Patients will be followed with MRI every 3 months (+/- 7 days) for the first year and then every 6 months (+/- 7 days) thereafter which is the standard of care.
  Arms: Cohort 2

SUMMARY:
The purpose of this study is to compare two different imaging methods to examine the response of brain metastases to WBRT. These two imaging methods will take pictures of the brain using : 1) a positron emission tomography (PET) scanner and 2) Magnetic Resonance Imaging (MRI) scanner. A PET scanner resembles a CT or MR scanner.PET scans use radioactive substances also called as radioactive markers to "see" cancer cells. We plan to use [18F]FLT as a radioactive marker. FLT is used to image tumor growth. FLT PET scan is a new clinical procedure. It is in the testing stage of development unlike FDG-PET which is used more commonly used. Therefore, this is considered a "research" study. This will help us evaluate whether this scan will be safe and better used in the future to evaluate tumors. The amount of radiation to the body is small. The radiation from the radiotracer drug will be gone from the body in a few hours. There is no radiation risk from the MRI scans. Additionally, we also plan to use MRI imaging of the brain. We expect that [18F]FLT PET is better when compared to MRI and will give us more information about the brain metastases after WBRT.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed (confirmation done at MSKCC) metastatic adenocarcinoma of the breast
* Radiologic evidence of new and/or progressive brain metastases ((≥10 mm in longest dimension) by MRI imaging of the Brain
* Planned WBRT based on number (≥ 3 lesions) and/or size (≥ 1 cm) of brain metastases.
* Age ≥18 years; males and females
* Patients who require additional clinically indicated stereotactic radiosurgery (SRS) in addition to WBRT will also be eligible.
* Life expectancy of >12 weeks.
* Karnofsky Performance Status (KPS) ≥ 70%.
* Creatinine ≤2.0 times the upper limit of normal.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to enrollment, must be non-lactating and must agree to use adequate contraception prior to enrollment and for the duration of study participation.
* No limit to prior therapies with last anti-cancer treatment ≥2 weeks from initiation of WBRT. Please note: there is no washout period required for trastuzumab, pertuzumab, for patients who have developed new parenchymal brain metastases while on these agents.

Exclusion Criteria:

* Leptomeningeal metastases Please note: leptomeningeal metastases may be allowed if it is limited to cranial metastasis (MRI spine should be completed, within 4 weeks of enrollment, to show that no other leptomeningeal metastases is present) and is not the only metastasis present in the brain.
* Concurrent administration of lapatinib or other tyrosine kinase inhibitors other than sorafenib
* Craniotomy or any other major surgery, open biopsy, or significant traumatic injury within 4 weeks of randomization.
* Concurrent anti-cancer therapy (chemotherapy, hormonal therapy, radiation therapy, surgery, immunotherapy, biologic therapy, or tumor embolization) other than sorafenib, and protocol-specified whole-brain radiotherapy.
* Use of any investigational drug within 30 days or 5 half-lives, whichever is longer, preceding enrollment.
* Inability to comply with protocol and /or not willing or not available for follow-up assessments.
* Any condition which in the investigator's opinion makes the patient unsuitable for the study participation.
* Patient is incontinent of urine or stool (which would make them unable to tolerate lying still for 60 minutes).
* Claustrophobia
* Known allergic reaction to Gd-DTPA
* Renal insufficiency with recent (<3 month old) creatinine >2.0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-06-13 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Seidman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York

REFERENCES:
- [Derived] Morikawa A, Grkovski M, Patil S, Jhaveri KL, Tang K, Humm JL, Holodny A, Beal K, Schoder H, Seidman AD. A phase I trial of sorafenib with whole brain radiotherapy (WBRT) in breast cancer patients with brain metastases and a correlative study of FLT-PET brain imaging. Breast Cancer Res Treat. 2021 Jul;188(2):415-425. doi: 10.1007/s10549-021-06209-4. Epub 2021 Jun 10. PMID 34109515
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: 12-039 is a companion FLT-PET brain imaging study to 12-046.
  10 participants from 12-046 were consented to 12-039. 10 other participants were approached for FLT-PET brain imaging getting standard WBRT off of 12-046, (without sorafenib), as a comparator group (not "arm").
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 12 | 5
Completed | 12 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 12-039 is a companion FLT-PET brain imaging study to 12-046.
Groups:
- Cohort 1: All participants will be imaged using FLT-PET scans at baseline (within 4 weeks of initiation of WBRT), 7-10 days after completion of WBRT and then 10-12 weeks after WBRT.
  Participants will also be evaluated with MRI imaging at baseline and then 10-12 weeks after WBRT.
  Participants will be followed with MRI every 3 months (+/- 7 days) for the first year and then every 6 months (+/- 7 days) thereafter which is the standard of care.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 12 | 5 | 17
Age, Continuous [Median (Full Range); unit: years] | 58 [43 to 77] | 53 [37 to 57] | 53 [37 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 0 | 11
  Male | 1 | 5 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 9 | 4 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 8 | 4 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall Response Rate is the proportion of participants who had a complete or partial response (Cohort 1)
Time Frame: 1 year
Population: 12-039 is a companion FLT-PET brain imaging study to 12-046.
  10 participants from 12-046 were consented to 12-039. 10 other participants were approached for FLT-PET brain imaging getting standard WBRT off of 12-046, (without sorafenib), as a comparator group (not "arm").
Measure: Number; unit: % of pts w/complete or partial response
Groups:
- Participants With Metastatic Breast Cancer: All participants will be imaged using FLT-PET scans at baseline (within 4 weeks of initiation of WBRT), 7-10 days after completion of WBRT and then 10-12 weeks after WBRT.
  Participants will also be evaluated with MRI imaging at baseline and then 10-12 weeks after WBRT.
  Participants will be followed with MRI every 3 months (+/- 7 days) for the first year and then every 6 months (+/- 7 days) thereafter which is the standard of care.
Arm/Group | Participants With Metastatic Breast Cancer
Number analyzed (Participants) | 12
% of pts w/complete or partial response | 71

2. Secondary Outcome: Change in Avg SUV Max From Baseline to 1 Year
Description: Comparing FLT PET findings with tissue analysis will enable us to determine if imaging results are concordant with histological findings and thus allow for confirmation of this hypothesis. In this manner, we propose to generate a bridge between tissue analysis and FLT-PET brain imaging studies. For patients needing to undergo craniotomy for resection of a brain metastasis after WBRT, tissue findings (radionecrosis versus viable tumor) will be correlated with radiologic assessment in an exploratory manner.
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Cohort 2: All participants will be imaged using FLT-PET scans at baseline (within 4 weeks of initiation of WBRT), 7-10 days after completion of WBRT and then 10-12 weeks after WBRT.
  Participants will also be evaluated with MRI imaging at baseline and then 10-12 weeks after WBRT.
  Participants will be followed with MRI every 3 months (+/- 7 days) for the first year and then every 6 months (+/- 7 days) thereafter which is the standard of care.
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 12 | 5
participants
  Not enrolled in FLT-PET study | 2 | 0
  Decline in avg SUV max of >/= 25% of WBRT + sorafenib participants | 9 | 0
  No decline in avg SUV max of >/= 25% of WBRT + sorafenib participants | 1 | 0
  Decline in avg SUV max of >/= 25% of WBRT participants | 0 | 2
  No decline in avg SUV max of >/= 25% of WBRT participants | 0 | 3

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Cohort 1: 12-039 is a companion FLT-PET brain imaging study to 12-046.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 10/12 | 5/5
Serious Adverse Events (participants affected / at risk) | 0/12 | 4/5
Other Adverse Events (participants affected / at risk) | 0/12 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=12) | Cohort 2 (N=5)
Blurred vision (Eye disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Lung Infection (Infections and infestations) | 0 | 1
Muscle weakness right-sided (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT01621906/Prot_SAP_000.pdf